CLINICAL TRIAL: NCT04784767
Title: Randomized Double-blind Placebo-Controlled Study in Healthy Adults to Evaluate Safety/Tolerability/Immunogenicity of Ranging Doses SARS-COV-2SPFN_1B-06-PL With Army Liposomal Formulation QS21 (ALFQ) for Prevention of COVID-19
Brief Title: PHASE 1 SARS-COV-2-Spike-Ferritin-Nanoparticle (SpFN) Vaccine With ALFQ Adjuvant for Prevention of COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: S-20-03; WRAIR # 2847 (Other: WRAIR); EID030 (Other: HJF); IND 27301 (Other: FDA)
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: SARS-CoV-2 Infection
Keywords: COVID-19; SARS-Cov-2; SARS; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — saponin QA-21V1; Sodium Chloride; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 1A: 25 µg of SpFN + ALFQ on Days 1, 29 and 181. (Experimental): Up to 20 participants will receive 25 µg of SpFN_1B-06-PL vaccine with 0.5 mL ALFQ adjuvant in a total 1.0 mL injection volume.
  Interventions: Biological: 25 µg SpFN_1B-06-PL + ALFQ (QS21 Adjuvant)
- 1B: Placebo (Sodium chloride, USP, for injection (0.9% NaCl) on Days 1, 29 and 181. (Placebo Comparator): 4 participants will receive 1.0mL of normal saline as Placebo on Study Days 1, 29, and 181.
  Interventions: Drug: Sodium chloride, USP, for injection (0.9% NaCl)
- 2A: 50 µg of SpFN + ALFQ on Days 1, 29, and 181. (Experimental): Up to 20 participants will receive 3 intramuscular injections of: 50 ug of SpFN_1B-06-PL with 0.5 mL ALFQ adjuvant.
  Interventions: Biological: 50 µg SpFN_1B-06-PL + ALFQ (QS21 Adjuvant)
- 2B: Placebo (Sodium chloride, USP, for injection (0.9% NaCl) on Days 1, 29, and 181. (Placebo Comparator): 4 participants will receive 1.0mL of normal saline as Placebo on Study Days 1, 29, and 181.
  Interventions: Drug: Sodium chloride, USP, for injection (0.9% NaCl)
- 3A: 50 µg of SpFN + ALFQ on Days 1 and 181. (Experimental): Up to 20 participants will receive 2 intramuscular injections of: 50 ug of SpFN_1B-06-PL with 0.5 mL ALFQ adjuvant.
  Interventions: Biological: 50 µg SpFN_1B-06-PL + ALFQ (QS21 Adjuvant)
- 3B: Placebo (Sodium chloride, USP, for injection (0.9% NaCl) on Days 1 and 181. (Placebo Comparator): 4 participants will receive 1.0mL of normal saline as Placebo on Study Days 1 and 181.
  Interventions: Drug: Sodium chloride, USP, for injection (0.9% NaCl)

INTERVENTIONS:
Biological: 25 µg SpFN_1B-06-PL + ALFQ (QS21 Adjuvant) — SpFN_1B-06-PL will be provided in a sterile, 2 mL single-use vial at 0.7 mL/vial, 90-110 ug/mL; ALFQ will be provided in a sterile 3 mL vial at 0.6 mL/vial
  Other Names: 25 µg SpFN + ALFQ
  Arms: 1A: 25 µg of SpFN + ALFQ on Days 1, 29 and 181.
Drug: Sodium chloride, USP, for injection (0.9% NaCl) — Normal saline will be provided in a sterile, single-use 10 mL vial
  Other Names: Placebo
  Arms: 1B: Placebo (Sodium chloride, USP, for injection (0.9% NaCl) on Days 1, 29 and 181.; 2B: Placebo (Sodium chloride, USP, for injection (0.9% NaCl) on Days 1, 29, and 181.; 3B: Placebo (Sodium chloride, USP, for injection (0.9% NaCl) on Days 1 and 181.
Biological: 50 µg SpFN_1B-06-PL + ALFQ (QS21 Adjuvant) — SpFN_1B-06-PL will be provided in a sterile, 2 mL single-use vial at 0.7 mL/vial, 90-110 ug/mL; ALFQ will be provided in a sterile 3 mL vial at 0.6 mL/vial
  Other Names: 50 µg SpFN + ALFQ
  Arms: 2A: 50 µg of SpFN + ALFQ on Days 1, 29, and 181.; 3A: 50 µg of SpFN + ALFQ on Days 1 and 181.

SUMMARY:
The purpose of this study is to evaluate the safety, reactogenicity, and immune response of the SpFN COVID-19 vaccine with Army Liposomal Formulation QS21 (ALFQ) adjuvant in healthy adults ages 18-55.

DETAILED DESCRIPTION:
This clinical protocol outlines a first-in-human study of the safety, tolerability, and immunogenicity of different doses of SpFN_1B-06-PL + ALFQ prophylactic vaccine against COVID-19 in healthy adults. The experimental vaccine in this study contains 2 parts: the vaccine (called SpFN_1B-06-PL) and an experimental adjuvant called ALFQ. An adjuvant is a substance added to vaccines that can help to make the vaccine more effective by improving the immune response or causing the immune response to last longer. The experimental vaccine in this study does not contain the virus and cannot cause you to become infected with the COVID-19 disease.

A total of 72 healthy adult participants (age range 18-55) will be enrolled in this study. Participants will be enrolled into one of three study arms:

Arm 1: 25 µg of SpFN_1B-06-PL vaccine with 0.5 mL ALFQ adjuvant in a total 1.0 mL injection volume (20 participants) or Placebo (4 participants) on Study Days 1, 29, and 181.

Arm 2: 50 µg of SpFN_1B-06-PL vaccine with 0.5 mL ALFQ adjuvant in a total 1.0 mL injection volume (20 participants) or Placebo (4 participants) on Study Days 1, 29, and 181.

Arm 3: 50 µg of SpFN_1B-06-PL vaccine with 0.5 mL ALFQ adjuvant in a total 1.0 mL injection volume (20 participants) or Placebo (4 participants) on Study Days 1 and 181.

Participants will:

* Be randomly assigned to get either the experimental COVID-19 vaccine or a placebo
* Receive 2 or 3 vaccine or placebo injections in the same arm muscle
* Record any side effects that they may experience for 7 days after receiving the injections.
* Have blood, nose swabs, and saliva samples collected at each visit.
* Have urine samples collected for pregnancy testing (females only).
* Undergo medical and physical examinations.
* Answer questions about potential exposures to COVID-19 in their daily life.

The duration of this study will be for about 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Must be a male or non-pregnant, non-breastfeeding female between the ages of 18 and 55 years, inclusive, at the time of enrollment.
* Must be willing and able to read, sign, and date the informed consent document.
* Must demonstrate an understanding of the study with a passing score (90% or greater) on the Test of Understanding (TOU) by the third attempt, before study-related procedures are performed.
* Must be willing and able to comply with study requirements and be available for follow-up visits for the entire study.
* Must have the means to be contacted by telephone and/or video for remote follow-up visits as needed.
* Must have a body mass index (BMI) ≥18.1 kg/m2 and <35.0 kg/m2.
* Have no previously documented COVID-19/SARS-CoV-2 infection
* Must agree to refrain from donating blood or plasma outside of this study for the duration of participation in this study.
* Must have acceptable screening laboratory findings: white blood cell (WBC), hemoglobin, platelet count, prothrombin (PT), prothrombin time (PTT), aspartate transaminase (AST), alanine transaminase (ALT), alkaline phosphatase (ALP), creatinine, and total bilirubin) within 14 days before Study Day 1.
* Must be healthy based on the physician investigator's clinical judgment after review of past medical history, medication use, vital signs, and an abbreviated physical examination.
* Biological females must have a negative urine pregnancy test at screening and a negative urine pregnancy test immediately before each study injection.
* Biological females of reproductive capacity must use an acceptable method of contraception, beginning 30 days before enrollment, and until at least 60 days after the last study injection.

Exclusion Criteria:

* Has plans to become pregnant or is currently pregnant or breastfeeding.
* Seropositive to COVID-19 by binding antibody titer assay.
* Confirmed positive for active infection of human immunodeficiency virus (HIV), hepatitis C virus (HCV), or presence of Hepatitis B surface antigen (HbsAg).
* Has known or suspected congenital or acquired immunodeficiency, or recent history or current use of immunosuppressive therapy.
* History of organ and or stem cell transplantation.
* Has a history of malignancy other than squamous cell or basal cell skin cancer, unless there has been surgical excision that is considered to have achieved a cure.
* Has diabetes mellitus type 1 or type 2 (including cases controlled with diet alone) and/or thyroid disease.
* Has major psychiatric illness during the last 12 months that, in the physician investigator's opinion, would preclude participation.
* Has a history of other chronic diseases or conditions
* Has a current or history of substance abuse that, in the physician investigator's opinion, would preclude participation.
* Has tattoos, scars, or other marks that would, in the opinion of the physician investigator, interfere with the assessment of the injection site.
* Has a known allergy or history of anaphylaxis or other serious reaction to a vaccine, vaccine component, or latex.
* Had major surgery (per the physician investigator's judgment) in the month before screening or has plans to have major surgery during the study.
* Received blood products or immunoglobulin in the three months before screening or has plans to use during the study.
* Donated a unit of blood within eight weeks before Study Day 1 or has plans to donate blood during the study.
* Received an experimental COVID-19 vaccine outside of this study or a COVID-19 vaccine that has been given Emergency Use Authorization from the FDA
* Received live attenuated vaccine from 30 days before Study Day 1 until 30 days after the last study injection.
* Received killed or inactivated vaccine from 14 days before Study Day 1 and until 30 days after the last study injection.
* Received experimental therapeutic agents within three months before the first study injection or has plans to receive any experimental therapeutic agents during the entire course of the study.
* Concurrent participation in another study requiring blood draws or exposure to investigational or non-investigational vaccine/product (pharmaceutical or device) throughout the study period.
* Has an acute illness or temperature ≥38.0 degrees Celsius (C)/100.4 degrees Fahrenheit (F) on any study injection day or within 48 hours of planned study injection.
* In the physician investigator's opinion, is unable to communicate reliably, is unlikely to adhere to study requirements, or has a condition that would limit completion of the study.
* Is unwilling to have their samples collected and stored for future research.
* Emergency medical services personnel and healthcare provider with patient contact in potentially high risk/high exposure settings as per screening physician's assessment.
* Current smoker or inhales vaporized nicotine "Vaping" daily. Current smoker is defined as an adult who has smoked 100 cigarettes in his or her lifetime and who currently smokes cigarettes.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with local and systemic reactions | Day 0 to 7 post vaccination
  Post-vaccination reactions including erythema, induration, pain/tenderness, swelling, limitation of arm movement, fever, tiredness, chills, rash, myalgia, arthralgia, nausea, and headache.
Incidents of treatment-adverse events as assessed by FDA Toxicity grading scale. | Day 0 to 546 post vaccination
  Number of participants with treatment related adverse events on Day 0 through day 546.
Number of participants with humoral immune response at Study Day 43 (+/- 2). | Day 43 (+/- 2 days)
  Number of participants with quantitative humoral immune response at Day 43, two weeks after the second SpFN_1B-06-PL + 0.5 mL ALFQ vaccine administration in Arms 1 & 2 and six weeks after the first administration in Arm 3.

SECONDARY OUTCOMES:
Number of participants with binding antibody response rate | Days 8, 15, 29, 43, and 57.
  The proportion of participants with detectable binding antibody responses, at baseline and at Study Days 8, 15, 29, 43, and 57.
Number of participants with neutralizing antibody response rate | Days 8, 15, 29, 43, and 57.
  The proportion of participants with neutralizing antibody titers (NAb) titers at ≥50% neutralization cutoff at the lowest level of dilution that optimizes interpretation at baseline and at Study Days 8, 15, 29, 43, and 57.
Number of participants with ACE-2 binding inhibition | Day 0 to 57 post vaccination
  The proportion of participants with ACE-2 binding inhibition following SpFN_1B-06-PL + ALFQ vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Scott, M.D., MPH, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- WRAIR Clinical Trials Center, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ober Shepherd BL, Scott PT, Hutter JN, Lee C, McCauley MD, Guzman I, Bryant C, McGuire S, Kennedy J, Chen WH, Hajduczki A, Mdluli T, Valencia-Ruiz A, Amare MF, Matyas GR, Rao M, Rolland M, Mascola JR, De Rosa SC, McElrath MJ, Montefiori DC, Serebryannyy L, McDermott AB, Peel SA, Collins ND, Joyce MG, Robb ML, Michael NL, Vasan S, Modjarrad K; EID-030 Study Group. SARS-CoV-2 recombinant spike ferritin nanoparticle vaccine adjuvanted with Army Liposome Formulation containing monophosphoryl lipid A and QS-21: a phase 1, randomised, double-blind, placebo-controlled, first-in-human clinical trial. Lancet Microbe. 2024 Jun;5(6):e581-e593. doi: 10.1016/S2666-5247(23)00410-X. Epub 2024 May 15. PMID 38761816

DOCUMENTS (1):
  • Informed Consent Form (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/67/NCT04784767/ICF_000.pdf